CLINICAL TRIAL: NCT06352138
Title: Phase III, Multicentre, Double-blind, Randomised, Parallel, Equivalence Clinical Trial to Assess Efficacy, Safety of Megalabs® Recombinant i/v Human Erythropoietin Compared to Epogen® in Anaemia in Patients With Chronic Kidney Disease
Brief Title: Comparative Study of Two Recombinant Human Erythropoietin Products in Chronic Kidney Disease Patients
Acronym: ENCASE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Megalabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENCASE
Record Dates: First submitted 2024-03-11; First posted 2024-04-08 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — Administration, Intravenous; Epoetin Alfa

STUDY DESIGN:
Intervention Model Description: multicentre, double-blind, randomised, parallel, equivalence trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epoetin alfa Megalabs® injectable in intravenous application. (Experimental): Epoetin alfa Megalabs, Human recombinant epoetin alfa
  Interventions: Biological: Experimental: Epoetin alfa Megalabs® Erythropoietin injectable in intravenous administration.
- Epoetin alfa Epogen® injectable in intravenous application. (Active Comparator): USA licenced Epoetin alfa, Epogen®, Human recombinant epoetin alfa
  Interventions: Biological: Active comparator: European Union licenced epoetin alfa

INTERVENTIONS:
Biological: Experimental: Epoetin alfa Megalabs® Erythropoietin injectable in intravenous administration. — comparison vs the reference product to demonstrate biological similarity
  Other Names: Epoetin alfa Megalabs®, Human recombinant epoetin alfa
  Arms: Epoetin alfa Megalabs® injectable in intravenous application.
Biological: Active comparator: European Union licenced epoetin alfa — comparison vs. the test product to demonstrate biological similarity
  Other Names: Epogen®, Human recombinant epoetin alfa
  Arms: Epoetin alfa Epogen® injectable in intravenous application.

SUMMARY:
Phase III, multicentre, double-blind, randomised, parallel, equivalence clinical trial to determine the efficacy, safety and immunogenicity of Megalabs® recombinant human alfa epoetin for intravenous use, compared to Epogen®, in the treatment of anaemia in participants with chronic renal disease, dependent on haemodialysis

DETAILED DESCRIPTION:
Patients with chronic kidney disease undergoing hemodialysis will be administered human recombinant alfa epoetin to revert anemia. Hemoglobin, hematocrit and reticulocyte counts will be assessed. Immunogenicity will be evaluated through bi-weekly Anti Drug Antibody determination. Test drug and comparator drug will be compared to evaluate biosimilarity.

ELIGIBILITY:
Inclusion Criteria:

* Stage V Chronic kidney disease undergoing hemodialysis

Exclusion Criteria:

* Lack of consent to participate in the trial, other severe chronic disease, history of pure red cell aplasia, existence of anti erythropoietin antibodies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Mean Absolute Change in Hemoglobin Levels | 18 months
  Response to epoetin alfa in patients with chronic kidney failure is an increase in hematocrit, hemoglobin and reduced transfusion requirements.
  Hemoglobin is the primary endpoint of the study .
Change in Mean Hb Level | 18 months
  Response to epoetin alfa in patients with chronic kidney failure is an increase in hematocrit, hemoglobin and reduced transfusion requirements.
  Hemoglobin is the primary endpoint of the study.

SECONDARY OUTCOMES:
immunogenicity | 18 months
  Anti-drug antibodies will be assessed in both groups every two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Kumar, MD, Study Director — Azidus Principal Investigator
Locations (1):
- Megalabs, Colonia Nicolich, Departamento de Canelones, Uruguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: reference guideline — https://www.ema.europa.eu/en/similar-biological-medicinal-products-containing-recombinant-erythropoietins-scientific-guideline